CLINICAL TRIAL: NCT01161407
Title: Calcium and Phosphorus Balance and Calcium Kinetics in Patients With Stage 3/4 Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Purdue University (Other)
Responsible Party: Principal Investigator, Munro Peacock, Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Genzyme - 0907-07
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Calcium; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo control for calcium carbonate, given in same capsule form as the calcium carbonate, 3 times per day with meals.
  Interventions: Dietary Supplement: Placebo
- Calcium Carbonate (Phosphate Binder) (Active Comparator): 500 mg elemental calcium as calcium carbonate given 3 times per day with meals for a total of 1500 mg/d elemental calcium.
  Interventions: Dietary Supplement: 1500 mg/d elemental calcium as calcium carbonate

INTERVENTIONS:
Dietary Supplement: 1500 mg/d elemental calcium as calcium carbonate — 500 mg elemental calcium as calcium carbonate given 3 times per day with meals for a total of 1500 mg/d elemental calcium. Given for 21 days in conjunction with a controlled diet.
  Arms: Calcium Carbonate (Phosphate Binder)
Dietary Supplement: Placebo — Placebo for calcium carbonate in same capsule form. Given 3 times per day with meals for 21 days in conjunction with a controlled diet.
  Arms: Placebo

SUMMARY:
The purpose of this study is to gain a better understanding of calcium absorption and metabolism in patients with Chronic Kidney Disease (CKD) using calcium balance and kinetic methods.

DETAILED DESCRIPTION:
The purpose of this study is to gain a better understanding of calcium absorption and metabolism in patients with Chronic Kidney Disease (CKD). It is important that the body get enough calcium to support many important body functions including bone health. CKD changes the calcium balance or how calcium is absorbed and excreted. Because of this, the knowledge of calcium absorption and excretion in patients with normal kidney function cannot be used to assess patients with CKD. In patients with CKD bone heath is often negatively affected due to a combination of poor calcium absorption, increased bone turnover (process where old bone is removed and new bone is formed), increased level of parathyroid hormone (PTH [ a hormone that acts to increase calcium in the blood]) and decrease in vitamin D levels. This negative effect is referred to as Chronic Kidney Disease Mineral Bone Disorder (CKD-MBD).

Treatment to correct CKD-MBD should begin early in the course of CKD. In the normal population calcium supplements are frequently used to help prevent age related bone loss. Calcium supplements can also be used in CKD patients to help bind phosphate. Maintaining correct levels of phosphate in the body is crucial in CKD. However, calcium supplements may have adverse effects by promoting calcium phosphate deposits in soft tissues like the vascular system which could increase the risk of cardiovascular disease.

Therefore this formal balance study is needed to determine if positive calcium balance occurs in patients with advanced CKD who are given calcium with meals as a phosphate binder. This study will also evaluate how the body handles phosphate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a GFR of < 45 ml/min;
2. Intact serum PTH > 37 pg/ml;
3. Age > 35 years (both genders and all races);
4. Able to perform two three-week balance studies;
5. Not on oral calcium or vitamin D other than multi vitamin, or willing to stop calcium or vitamin D for one month prior to entry in the study (day 1 of first calcium balance period);
6. Female patients must be post-menopausal (defined as last menstrual period at least 12 months prior to screening visit) or surgically sterile by hysterectomy;
7. On stable doses of diuretics, bisphosphonates, anti-epileptics (except dilantin) for at least 2 months.

Exclusion Criteria:

1. Serious underlying systemic disease (including uncontrolled diabetes, lupus, hypertension, amyloid, etc);
2. Taking drugs that alter calcium and phosphate balance or homeostasis including high dose cholecalciferol or ergocalciferol (1000 U/day or 50,000U/ wk, respectively), active vitamin D metabolites, calcimimetics, PTH analogues in the last 30 days;
3. Taking drugs that the investigator feels will alter calcium balance;
4. Plan to initiate dialysis in the next six months;
5. Hypercalcemia defined as serum calcium > 10.5 mg/dl;
6. Hyperphosphatemia defined as serum phosphate >5.5mg/ml;
7. Intestinal disease that alters absorption or normal intestinal function including celiac disease, small bowel resection, bariatric surgery;
8. Smoking

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Munro Peacock, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital - Clinical Research Center, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Francis RM, Peacock M, Barkworth SA. Renal impairment and its effects on calcium metabolism in elderly women. Age Ageing. 1984 Jan;13(1):14-20. doi: 10.1093/ageing/13.1.14. PMID 6422710
- [Background] Levin A, Bakris GL, Molitch M, Smulders M, Tian J, Williams LA, Andress DL. Prevalence of abnormal serum vitamin D, PTH, calcium, and phosphorus in patients with chronic kidney disease: results of the study to evaluate early kidney disease. Kidney Int. 2007 Jan;71(1):31-8. doi: 10.1038/sj.ki.5002009. Epub 2006 Nov 8. PMID 17091124
- [Background] Kestenbaum B, Sampson JN, Rudser KD, Patterson DJ, Seliger SL, Young B, Sherrard DJ, Andress DL. Serum phosphate levels and mortality risk among people with chronic kidney disease. J Am Soc Nephrol. 2005 Feb;16(2):520-8. doi: 10.1681/ASN.2004070602. Epub 2004 Dec 22. PMID 15615819
- [Background] Jackman LA, Millane SS, Martin BR, Wood OB, McCabe GP, Peacock M, Weaver CM. Calcium retention in relation to calcium intake and postmenarcheal age in adolescent females. Am J Clin Nutr. 1997 Aug;66(2):327-333. doi: 10.1093/ajcn/66.2.327. PMID 9250111
- [Background] Coburn JW, Hartenbower DL, Massry SG. Intestinal absorption of calcium and the effect of renal insufficiency. Kidney Int. 1973 Aug;4(2):96-104. doi: 10.1038/ki.1973.88. No abstract available. PMID 4275344
- [Background] Peacock M, Aaron JE, Walker GS, Davison AM. Bone disease and hyperparathyroidism in chronic renal failure: the effect of 1alpha-hydroxyvitamin D3. Clin Endocrinol (Oxf). 1977 Dec;7 Suppl:73s-81s. doi: 10.1111/j.1365-2265.1977.tb03365.x. No abstract available. PMID 606428
- [Background] Weaver CM, Martin BR, Plawecki KL, Peacock M, Wood OB, Smith DL, Wastney ME. Differences in calcium metabolism between adolescent and adult females. Am J Clin Nutr. 1995 Mar;61(3):577-81. doi: 10.1093/ajcn/61.3.577. PMID 7872222
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Stremke ER, McCabe LD, McCabe GP, Martin BR, Moe SM, Weaver CM, Peacock M, Hill Gallant KM. Twenty-Four-Hour Urine Phosphorus as a Biomarker of Dietary Phosphorus Intake and Absorption in CKD: A Secondary Analysis from a Controlled Diet Balance Study. Clin J Am Soc Nephrol. 2018 Jul 6;13(7):1002-1012. doi: 10.2215/CJN.00390118. Epub 2018 Jun 19. PMID 29921736
- [Derived] Hill KM, Martin BR, Wastney ME, McCabe GP, Moe SM, Weaver CM, Peacock M. Oral calcium carbonate affects calcium but not phosphorus balance in stage 3-4 chronic kidney disease. Kidney Int. 2013 May;83(5):959-66. doi: 10.1038/ki.2012.403. Epub 2012 Dec 19. PMID 23254903
- See also: Pubmed entry of publication from this study. — http://www.ncbi.nlm.nih.gov/pubmed/23254903

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcium Then Placebo: Crossover order was calcium then placebo, separated by at least a 3 week washout period.
  Calcium treatment was 1500 mg/d calcium as calcium carbonate given as three 500 mg calcium capsules at each of the three meals per day. Placebo was identical in shape, appearance, and administration.
- Placebo Then Calcium: Crossover order was placebo then calcium, separated by at least a 3 week washout period.
  Calcium treatment was 1500 mg/d calcium as calcium carbonate given as three 500 mg calcium capsules at each of the three meals per day. Placebo was identical in shape, appearance, and administration.
Period: Overall Study
Arm/Group | Calcium Then Placebo | Placebo Then Calcium
Started | 6 | 6
Completed | 3 | 5
Not Completed | 3 | 1
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium Then Placebo | Placebo Then Calcium | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (8.1) | 60.8 (5.3) | 57.4 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Calcium Balance
Description: Calcium balance is measured by dietary calcium intake (mg/d) minus calcium excretion (mg/d) (from both urine and feces).
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/d calcium
Arm/Group | Placebo | Calcium
Number analyzed (Participants) | 8 | 8
mg/d calcium | 61 (60) | 508 (60)

2. Secondary Outcome: Phosphorus Balance
Description: Phosphorus balance is measured by dietary phosphorus intake (mg/d) minus phosphorus excretion (mg/d) from both urine and feces.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/d phosphorus
Arm/Group | Placebo | Calcium
Number analyzed (Participants) | 8 | 8
mg/d phosphorus | 95 (29) | 153 (29)

3. Secondary Outcome: "Bone Balance" From Calcium Kinetics
Description: Calcium kinetics was determined by a calcium radiotracer. Bone balance is the difference between bone formation and bone resorption estimated by calcium kinetic modeling.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/d calcium
Arm/Group | Placebo | Calcium
Number analyzed (Participants) | 8 | 8
mg/d calcium | 62 (42) | 259 (42)

ADVERSE EVENTS:
Arm/Group | Placebo | Calcium
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Due to the characteristic short treatment periods of balance studies, the results may not reflect the effects of chronic treatment with calcium carbonate on mineral balance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days